CLINICAL TRIAL: NCT03669133
Title: Vitamin E for NASH Treatment in HIV Infected Individuals
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of coordinator resources and lack of access to study resources during and due to the COVID pandemic
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Samer Gawrieh, Associate Professor of Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1807274844
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: NAFLD; NASH - Nonalcoholic Steatohepatitis; HIV Infections
Keywords: Fatty liver; NAFLD; NASH; HIV; Vitamin E
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; HIV Infections; Fatty Liver | interventions — Vitamin E

STUDY DESIGN:
Intervention Model Description: Group A: Vitamin E 800 IU/daily for 24 weeks. (total of 28 subjects) Group B: Matching placebo for 24 weeks (total of 28 subjects)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study biostatistician and Investigational Drug Services pharmacist will randomize subjects and will provide study drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Vitamin E 800 IU/daily for 24 weeks
  Interventions: Drug: Vitamin E
- Group B (Placebo Comparator): Matching placebo for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin E — Vitamin E 800 IU/daily
  Arms: Group A
Drug: Placebo — Matching placebo daily
  Arms: Group B

SUMMARY:
The purpose of this study is to see how taking Vitamin E daily affects fatty liver in persons living with HIV. Subjects will have both HIV and a fatty liver and the purpose of the study is to learn if underlying liver condition (fatty liver) gets better, worse, or stays the same from taking Vitamin E.

DETAILED DESCRIPTION:
The investigators will conduct a proof-of-concept clinical trial to evaluate the efficacy of vitamin E for treatment of non-alcoholic steatohepatitis (NASH) in persons living with HIV. Hypothesis: Vitamin E will improve radiographically measured hepatic fat content and circulating markers of liver inflammation and injury in persons living with HIV who have NASH.

A. Perform a pilot randomized placebo controlled trial of vitamin E 800 IU/daily for 6 months in 56 persons living with HIV with biopsy-proven NASH B. Measure change in liver fat content by magnetic resonance proton-density fat fraction (Primary outcome) C. Determine the impact of vitamin E treatment on noninvasive markers of hepatic and systemic inflammation, hepatic fibrosis, and systemic oxidative stress (Secondary outcomes) D. Define baseline hepatic gene expression signatures predictive of response to therapy.

Upon completion, the proposed clinical trial may establish vitamin E as an excellent and inexpensive candidate for further development as a treatment for NASH in persons living with HIV.

ELIGIBILITY:
Inclusion Criteria:

1. males and females ≥18 years with biopsy-proven NASH within 6 months prior to enrollment
2. histological diagnosis of NASH will be confirmed by an experienced liver pathologist before study entry
3. HIV infection
4. stable dose of anti-diabetic agents and ART in the 3 months preceding enrollment and expected by the physician treating diabetes and HIV to remain on stable medications during the study
5. willingness to participate in the study
6. ability to understand and give informed consent for participation

Exclusion Criteria:

1. Presence of other chronic liver diseases (hepatitis B or C, autoimmune hepatitis, cholestatic liver disease, Wilson disease, hemochromatosis, etc.)
2. average alcohol consumption >3 drinks/day for men or >2 drinks/day for women in the 6 months prior to enrollment.
3. Alcohol Use Disorder Identification Test (AUDIT) score of ≥8
4. evidence of cirrhosis on histology or imaging
5. ongoing use of medications known to cause hepatic steatosis (e.g., corticosteroids, amiodarone, methotrexate, tetracycline, tamoxifen, estrogens at doses greater than those used for birth control, anabolic steroids, or valproic acid)
6. prior bariatric surgery
7. severe co-morbidities (e.g., advanced cardiac, renal, pulmonary, or psychiatric illness)
8. allergy to vitamin E
9. use of vitamin E or multivitamins containing vitamin E in the three months preceding enrollment
10. use of drugs with potential effect on NASH such as ursodeoxycholic acid, S-adenosylmethionine (SAM-e), betaine, pentoxifylline, or milk thistle in the three months prior to enrollment.
11. changing doses of statins (simvastatin, pravastatin, atorvastatin, fluvastatin, lovastatin, rosuvastatin) or fibrates (clofibrate, fenofibrate) in the three months prior enrollment.
12. illicit substance abuse within the past twelve months
13. breast feeding, pregnancy, inability or unwillingness to practice contraception for the duration of the study
14. contraindications for the MRI procedure (e.g., prostheses, severe claustrophobia)
15. poorly controlled diabetes with A1C >8.5 within in the last six months
16. use of total parenteral nutrition in the 6 months preceding liver biopsy or enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants consented to participate in this trial. One person screen-failed and two completed the trial, with one randomized to each arm.
Groups:
- Vitamin E 800 I/U: Vitamin E 800 I/U daily for 24 weeks
  Vitamin E: Vitamin E 800 I/U daily
- Placebo: Matching placebo for 24 weeks
  Placebos: Matching placebo daily
Period: Overall Study
Arm/Group | Vitamin E 800 I/U | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Three people consented to enroll in this study; one participant screen failed and two completed the study
Groups:
- Group B: Matching placebo for 24 weeks
  Placebos: Matching placebo daily
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (8.49) | 38 (8.49) | 44 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Liver Fat Content by Magnetic Resonance Proton-Density Fat Fraction
Description: change in liver steatosis via MRI-PDFF at randomization (day 1) and study completion (week 24) to assess liver steatosis
Time Frame: at randomization visit (study day 1) and end of study visit (week 24)
Population: change in liver steatosis via MRI-PDFF or the one participant in each group
Measure: Number; unit: percentage change
Groups:
- Vitamin E 800 I/U: Vitamin E 800 IU/daily for 24 weeks
  Vitamin E: Vitamin E 800 IU/daily
Arm/Group | Vitamin E 800 I/U | Placebo
Number analyzed (Participants) | 1 | 1
percentage change | 0 | 4

2. Secondary Outcome: Impact of Vitamin E Treatment on Noninvasive Markers of Hepatic Fibrosis
Description: This outcome measure reflects the change in liver stiffness in transient elastrography via FibroScan is measured in (kPa) for study participants at two study time points
Time Frame: change from baseline (first screening visit) to the end of study visit (week 24)
Population: Change in liver stiffness (LSM) via FibroScan for the one participant in each group
Measure: Number; unit: kPa - kilopascels
Arm/Group | Vitamin E 800 I/U | Placebo
Number analyzed (Participants) | 1 | 1
kPa - kilopascels | -28.3 | -0.8

3. Secondary Outcome: Impact of Treatment on ALT as a Noninvasive Marker of Hepatic Inflammation
Description: This measure reflects the change in ALT(IU/L) value for study participants at two study time points
Time Frame: at randomization visit (study day 1) and end of study visit (week 24)
Population: Change in ALT from study randomization (day 1) through the end of study visit (week 24)
Measure: Number; unit: IU/L
Arm/Group | Vitamin E 800 I/U | Placebo
Number analyzed (Participants) | 1 | 1
IU/L | -10 | 3

4. Secondary Outcome: Impact of Treatment on AST as a Noninvasive Marker of Hepatic Inflammation
Description: This measure reflects the change in AST(IU/L) value for study participants at two study time points
Time Frame: Change in AST from study randomization (day 1) through the end of study visit (week 24)
Population: one participant completed each group
Measure: Number; unit: IU/L
Arm/Group | Vitamin E 800 I/U | Placebo
Number analyzed (Participants) | 1 | 1
IU/L | -16 | 14

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment until the end of the study, for a total of 28 weeks.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=1) | Group B (N=1)
COVID (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Both participants, during the course of the study, contracted COVID.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03669133/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03669133/SAP_003.pdf